CLINICAL TRIAL: NCT00265902
Title: Ultra-Sensitive, Infra-Red Thermographic Analysis of Kaposi's Sarcoma Skin Lesions
Brief Title: Infrared Thermography in Finding Skin Lesions in Patients With Kaposi's Sarcoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: J0429; CDR0000452799 (Registry Identifier: PDQ (Physician Data Query)); JHOC-0429; 04-08-06-02 (Other: JHM IRB)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2006-06

CONDITIONS: Sarcoma
Keywords: Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Kaposi | interventions — X-Rays

INTERVENTIONS:
Procedure: diagnostic imaging

SUMMARY:
RATIONALE: Diagnostic procedures, such as infrared thermography, may help find Kaposi's sarcoma and learn the extent of disease.

PURPOSE: This clinical trial is studying how well infrared thermography finds skin lesions in patients with Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare ultra-sensitive infrared thermographic images with visible light digital photographic images and clinical dermatologic examination as methods of measuring cutaneous lesions in patients with Kaposi's sarcoma (KS).

Secondary

* Compare differences in modulation of temperature detected in KS skin lesions with non-involved skin of the same patient and with normal skin of healthy volunteers by sequential imaging using the infrared thermographic camera.

OUTLINE: This is a controlled, pilot study.

Patients undergo clinical assessment followed by simultaneous digital photographic camera imaging and high-resolution infrared thermographic camera imaging of designated normal skin areas and selected marker lesions. Before imaging, a metal bar chilled to 0º C, 10º C, and 25º C is applied to the lesions and designated normal skin areas for up to 90 seconds.

Healthy volunteers (controls) undergo the same procedure as for the patient except only designated normal skin areas are used.

PROJECTED ACCRUAL: A total of 20 patients and 10 healthy volunteers (controls) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Histologically confirmed cutaneous Kaposi's sarcoma (KS)

    * At least one skin lesion accessible for imaging
    * HIV positivity with proven cutaneous KS and concurrent visceral or mucous membrane involvement allowed
  * Healthy volunteer (regardless of HIV status) (control)

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Pregnancy allowed

PRIOR CONCURRENT THERAPY:

* Prior topical, intralesional, or systemic treatment allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-10-03 (Actual); Primary Completion 2006-03-21 (Actual); Study Completion 2006-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Martins, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States